CLINICAL TRIAL: NCT00186459
Title: GCRC-CAP-Tracey McLaughlin, MD
Brief Title: Obesity, Weight Loss, and Cardiovascular Disease Risk
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Tracey McLaughlin, Associate Professor, Stanford University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: RR16071-01
Record Dates: First submitted 2005-09-13; First posted 2005-09-16 (Estimated); Last update posted 2024-12-04 (Actual); Status verified 2024-12

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

INTERVENTIONS:
Behavioral: Hypocaloric diet of varying macronutrient composition

SUMMARY:
The goal of the study is to define the roles played by resistance to insulin-mediated glucose disposal (insulin resistance) and circulating plasma insulin concentrations in: 1) ability to lose weight; 2) reduction of risk for coronary heart disease as a result of weight loss. We hypothesize that in the setting of caloric restriction, manipulating endogenous insulin concentrations will not alter ability of subjects to lose weight, but will lead to different reduction in CHD risk factors. To test this hypothesis, two parallel studs will be performed. First, obese insulin-resistant individuals will be randomized to one of two equally-hypocaloric diets that vary moderately in proportion of carbohydrate and mono/polyunsaturated fats (lower carbohydrate diet will be associated with greater reduction in endogenous insulin secretion). Second, diabetics treated with insulin secretagogues will be compared to diabetics treated with insulin sensitizers with respect to the same outcomes (secretagogues increase insulin secretion and insulin sensitizers decrease insulin concentrations). Endpoints include weight loss, change in insulin resistance, blood pressure, lipid and lipoproteins, markers of endothelial function, daylong insulin and glucose concentrations: these will be compared, in each of the parallel studies, between the group with insulin-stimulating intervention vs the group with the insulin-sparing intervention.

DETAILED DESCRIPTION:
While obesity, insulin resistance, and diabetes are highly associated, it is not clear whether insulin resistance and compensatory hyperinsulinemia play important roles in the tendency to gain weight and/or inability to lose weight. The role of hyperinsulinemia in coronary heart disease (CHD)is also unclear. The specific aims of the proposed research are as follows:

1. To compare insulin resistant versus insulin sensitive nondiabetic overweight individuals with respect to their ability to lose weight on a low calorie diet. CHD risk factors before and after weight loss will also be assessed to determine the degree to which insulin resistance is associated with CHD risk, as well as the impact that differences in insulin resistance have on the metabolic benefits of weight loss
2. To determine if weight loss and its associated metabolic benefits vary as a function of the relative amounts of dietary fat and carbohydrate in hypocaloric diets. Because high carbohydrate diets increase insulin secretion, the relationship between dietary composition and change in circulating insulin concentrations will be analyzed with respect to both weight loss and CHD risk factors.
3. To quantify and compare the improvement in glycemic control and CHD risk factors associated with weight loss in obese type 2 diabetics, while being treated with 1) an insulin secretagogue (sulfonylurea) or 2) an insulin sensitizer (thiazolidinedione). Manipulation of plasma insulin concentrations with these medications will provide a mechanism by which to evaluate the impact of circulating insulin concentrations on the described outcome measures.
4. A subgroup of overweight/obese premenopausal women with PCOS will be studied using two diets in crossover design with regard to macronutrient effects on endogenous hyperinsulinism. For this subgroup age range will be 18-50 years, BMI 25-50 kg/m2.
5. In order to increase our data and therefore increase our better understanding of fat cells and insulin resistance and changes in fat cells with weight loss we would like to increase our participant enrollment to 550 all to be enrolled at Stanford University Medical Center recruiting Bariatric participants:

Age for Bariatric patients 30-65 men and women BMI 27-no upper limit Currently we have completed all participants except the bariatric and post bariatric population and those with hypoglycemia following bariatric surgery.

The ethnic background of subjects reflects Stanford's patient population.

ELIGIBILITY:
Inclusion Criteria:

* BMI 30-35
* age 35-65
* nondiabetic by fasting plasma glucose concentration
* no active major organ diseases
* insulin resistant or insulin sensitive

Exclusion Criteria:

* anemia
* pregnant
* major organ disease
* active malignancy
* eating disorder
* active psychiatric illness
* chronic inflammatory conditions

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2000-10; Primary Completion 2017-08-31 (Actual); Study Completion 2017-08-31 (Actual)

PRIMARY OUTCOMES:
Weight loss

SECONDARY OUTCOMES:
Lipid/lipoprotein changes
Blood pressure changes
Insulin resistance changes
Endothelial function changes

CONTACTS AND LOCATIONS:
Overall Officials: Dr Tracey Lynn McLaughlin, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States

REFERENCES:
- [Derived] McLaughlin T, Abbasi F, Lamendola C, Yee G, Carter S, Cushman SW. Dietary weight loss in insulin-resistant non-obese humans: Metabolic benefits and relationship to adipose cell size. Nutr Metab Cardiovasc Dis. 2019 Jan;29(1):62-68. doi: 10.1016/j.numecd.2018.09.014. Epub 2018 Oct 11. PMID 30497926
- [Derived] Perelman D, Coghlan N, Lamendola C, Carter S, Abbasi F, McLaughlin T. Substituting poly- and mono-unsaturated fat for dietary carbohydrate reduces hyperinsulinemia in women with polycystic ovary syndrome. Gynecol Endocrinol. 2017 Apr;33(4):324-327. doi: 10.1080/09513590.2016.1259407. Epub 2016 Dec 2. PMID 27910718